CLINICAL TRIAL: NCT00071487
Title: A Phase 2, Multi-Center, Double-Blind, Placebo-Controlled, Dose-Ranging Study to Evaluate the Safety, Tolerability, and Efficacy of LymphoStat-B™ Antibody (Monoclonal Anti-BLyS Antibody) in Subjects With Systemic Lupus Erythematosus (SLE)
Brief Title: Safety and Efficacy Study of LymphoStat-B (Belimumab) in Subjects With Systemic Lupus Erythematosus (SLE)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Human Genome Sciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LBSL02
Record Dates: First submitted 2003-10-24; First posted 2003-10-28 (Estimated); Results first posted 2012-08-28 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-08

CONDITIONS: Lupus Erythematosus, Systemic
Keywords: SLE
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — belimumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo plus SOC (Placebo Comparator)
  Interventions: Drug: Placebo
- Belimumab 1 mg/kg plus SOC (Experimental)
  Interventions: Drug: Belimumab 1 mg/kg
- Belimumab 4 mg/kg plus SOC (Experimental)
  Interventions: Drug: Belimumab 4 mg/kg
- Belimumab 10 mg/kg plus SOC (Experimental)
  Interventions: Drug: Belimumab 10 mg/kg

INTERVENTIONS:
Drug: Placebo — Placebo IV plus standard therapy (SOC) for SLE; placebo administered on Days 0, 14, 28, and every 28 days thereafter through 52 weeks in the double-blind period. In the open-label extension period, placebo patients who opted to participate received belimumab 10 mg/kg IV plus SOC every 28 days for an additional 24 weeks.
  Arms: Placebo plus SOC
Drug: Belimumab 1 mg/kg — Belimumab 1 mg/kg IV plus standard therapy (SOC) for SLE; belimumab 1 mg/kg administered on Days 0, 14, 28, and every 28 days thereafter through 52 weeks in the double-blind period. In the open-label extension period, patients who opted to participate either continued on the same dose of belimumab or may have been switched to belimumab 10 mg/kg at the investigator's discretion for an additional 24 weeks.
  Other Names: LymphoStat-B®; BENLYSTA®
  Arms: Belimumab 1 mg/kg plus SOC
Drug: Belimumab 4 mg/kg — Belimumab 4 mg/kg IV plus standard therapy (SOC) for SLE; belimumab 4 mg/kg administered on Days 0, 14, 28, and every 28 days thereafter through 52 weeks in the double-blind period. In the open-label extension period, patients who opted to participate either continued on the same dose of belimumab or may have been switched to belimumab 10 mg/kg at the investigator's discretion for an additional 24 weeks.
  Other Names: LymphoStat-B®; BENLYSTA®
  Arms: Belimumab 4 mg/kg plus SOC
Drug: Belimumab 10 mg/kg — Belimumab 10 mg/kg IV plus standard therapy (SOC) for SLE; belimumab 10 mg/kg administered on Days 0, 14, 28, and every 28 days thereafter through 52 weeks in the double-blind period. In the open-label extension period, patients who opted to participate continued on belimumab 10 mg/kg for an additional 24 weeks.
  Other Names: LymphoStat-B®; BENLYSTA®
  Arms: Belimumab 10 mg/kg plus SOC

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of 3 different doses of belimumab, administered in addition to standard therapy, in patients with active SLE disease.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety and efficacy of three different doses of belimumab (1 mg/kg, 4 mg/kg, and 10 mg/kg), administered in addition to standard therapy, compared to placebo plus standard therapy in patients with active SLE disease. Patients were randomly assigned, following stratification by the screening SELENA SLEDAI score (4 to 7 versus ≥ 8), to 1 of the 4 study arms (3 active arms and 1 placebo arm plus standard therapy for SLE). All patients were to be dosed on Days 0, 14, and 28, then every 28 days for the remainder of 52 weeks. Patients completing the 52-week period could enter a 24-week open-label extension; belimumab patients received the same dose or were switched to 10 mg/kg at the investigator's discretion and former placebo patients received belimumab 10 mg/kg.

ELIGIBILITY:
Primary Inclusion Criteria

* Clinical diagnosis of SLE
* "Active" SLE disease
* On a stable SLE treatment regimen
* History of measurable autoantibodies

Primary Exclusion Criteria

* Received a non-FDA approved investigational agent within last 28 days
* Cyclosporin, intravenous immunoglobulin (IVIG) or plasmapheresis within last 90 days
* Active lupus nephritis requiring hemodialysis, cyclophosphamide (Cytoxan™), or high-dose prednisone (> 100 mg/day) within last 90 days
* Active central nervous system (CNS) lupus requiring therapeutic intervention within last 60 days
* History of renal transplant
* History of chronic infection that has been active within last 6 months, herpes zoster within last 90 days or any infection requiring hospitalization or intravenous medication within last 60 days
* History of hypogammaglobulinemia or immunoglobulin A (IgA) deficiency
* Human immunodeficiency virus (HIV), Hepatitis B, Hepatitis C

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 449 (Actual)
Dates: Start 2003-10; Primary Completion 2005-08 (Actual); Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (62):
- United States (60):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Arizona Arthritis Research, Paradise Valley, Arizona
  - University of Arizona, Tucson, Arizona
  - Scripps Clinic, La Jolla, California
  - University of Southern California, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Stanford University School of Medicine, Palo Alto, California
  - Boling Clinical Trials, Rancho Cucamonga, California
  - UCDMC, Sacramento, California
  - Arthritis Care Center, Inc., San Jose, California
  - Arthritis Associates & Osteoporosis Center Of Colorado Springs, Colorado Springs, Colorado
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Arthritis and Rheumatic Disease Specialties, Aventura, Florida
  - Rheumatology Associates of Central Florida, Orlando, Florida
  - Tampa Medical Group, P.A., Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Radiant Research Boise, Boise, Idaho
  - Institute of Arthritis and Research, Idaho Falls, Idaho
  - Northwestern University Medical School, Chicago, Illinois
  - Rheumatology Associates, Chicago, Illinois
  - Medical Specialists, Munster, Indiana
  - Kentuckiana Center for Better Bone and Joint Health, Louisville, Kentucky
  - Ochsner Clinic Foundation, Baton Rouge, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - University of Maryland, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland
  - The Osteoporosis and Arthritis Clinical Trial Center, Cumberland, Maryland
  - Center for Rheumatology and Bone Research, Wheaton, Maryland
  - Tufts--New England Medical Center, Boston, Massachusetts
  - The University of Michigan Health System, Ann Arbor, Michigan
  - Washington University in St. Louis, St Louis, Missouri
  - Arthritis Center of Nebraska, Lincoln, Nebraska
  - Arthritis and Osteoporosis Center, Concord, New Hampshire
  - Strafford Medical Associates, P.A., Dover, New Hampshire
  - The Center for Rheumatology, Albany, New York
  - SUNY-Downstate Medical Center, Brooklyn, New York
  - North Shore University Hospital, Manhasset, New York
  - Aair Research, Rochester, New York
  - Jacobi Medical Center, The Bronx, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Arthritis Clinic and Carolina Bone and Joint, Charlotte, North Carolina
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - Stat Research Inc., Dayton, Ohio
  - Bone and Joint Hospital, Oklahoma City, Oklahoma
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - Oklahoma Center For Arthritis Therapy & Research, Tulsa, Oklahoma
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh School of Medicine & ASPH, Pittsburgh, Pennsylvania
  - Rheumatic Disease Associates, Willow Grove, Pennsylvania
  - Research Associates of North Texas, Dallas, Texas
  - UT Southwestern Medical Center at Dallas, Dallas, Texas
  - Texas Research Center, Sugar Land, Texas
  - Arthritis and Rheumatic Disease Clinic, Ogden, Utah
  - Physicians Research Options, LC, Sandy City, Utah
  - Arthritis Clinic of Northern Virginia, P.C., Arlington, Virginia
  - Edmonds Rheumatology Associates, Edmonds, Washington
  - Arthritis Northwest Rheumatology, Spokane, Washington
  - Gundersen Clinic, Ltd., La Crosse, Wisconsin
  - The Medical College of Wisconsin , Inc, Milwaukee, Wisconsin
  - Marshfield Medical Research Foundation, Wausau, Wisconsin
- Canada (2):
  - Toronto Western Hospital, Toronto, Ontario
  - McGill University Health Center, Montreal, Quebec

REFERENCES:
- [Result] Wallace DJ, Stohl W, Furie RA, Lisse JR, McKay JD, Merrill JT, Petri MA, Ginzler EM, Chatham WW, McCune WJ, Fernandez V, Chevrier MR, Zhong ZJ, Freimuth WW. A phase II, randomized, double-blind, placebo-controlled, dose-ranging study of belimumab in patients with active systemic lupus erythematosus. Arthritis Rheum. 2009 Sep 15;61(9):1168-78. doi: 10.1002/art.24699. PMID 19714604
- [Result] Furie RA, Petri MA, Wallace DJ, Ginzler EM, Merrill JT, Stohl W, Chatham WW, Strand V, Weinstein A, Chevrier MR, Zhong ZJ, Freimuth WW. Novel evidence-based systemic lupus erythematosus responder index. Arthritis Rheum. 2009 Sep 15;61(9):1143-51. doi: 10.1002/art.24698. PMID 19714615
- [Derived] Arends EJ, Zlei M, Tipton CM, Cotic J, Osmani Z, de Bie FJ, Kamerling SWA, van Maurik A, Dimelow R, Gregan YI, Fox NL, Rabelink TJ, Roth DA, Sanz I, van Dongen JJM, van Kooten C, Teng YKO. Disruption of memory B-cell trafficking by belimumab in patients with systemic lupus erythematosus. Rheumatology (Oxford). 2024 Sep 1;63(9):2387-2398. doi: 10.1093/rheumatology/keae286. PMID 38775637
- [Derived] Gupta SV, Fanget MC, MacLauchlin C, Clausen VA, Li J, Cloutier D, Shen L, Robbie GJ, Mogalian E. Clinical and Preclinical Single-Dose Pharmacokinetics of VIR-2218, an RNAi Therapeutic Targeting HBV Infection. Drugs R D. 2021 Dec;21(4):455-465. doi: 10.1007/s40268-021-00369-w. Epub 2021 Nov 6. PMID 34741731
- [Derived] Zhou X, Lee TI, Zhu M, Ma P. Prediction of Belimumab Pharmacokinetics in Chinese Pediatric Patients with Systemic Lupus Erythematosus. Drugs R D. 2021 Dec;21(4):407-417. doi: 10.1007/s40268-021-00363-2. Epub 2021 Oct 9. PMID 34628605
- [Derived] Brunner HI, Abud-Mendoza C, Mori M, Pilkington CA, Syed R, Takei S, Viola DO, Furie RA, Navarra S, Zhang F, Bass DL, Eriksson G, Hammer AE, Ji BN, Okily M, Roth DA, Quasny H, Ruperto N. Efficacy and safety of belimumab in paediatric and adult patients with systemic lupus erythematosus: an across-study comparison. RMD Open. 2021 Sep;7(3):e001747. doi: 10.1136/rmdopen-2021-001747. PMID 34531304
- [Derived] Hannon CW, McCourt C, Lima HC, Chen S, Bennett C. Interventions for cutaneous disease in systemic lupus erythematosus. Cochrane Database Syst Rev. 2021 Mar 9;3(3):CD007478. doi: 10.1002/14651858.CD007478.pub2. PMID 33687069
- [Derived] Ginzler EM, Wallace DJ, Merrill JT, Furie RA, Stohl W, Chatham WW, Weinstein A, McKay JD, McCune WJ, Zhong ZJ, Freimuth WW, Petri MA; LBSL02/99 Study Group. Disease control and safety of belimumab plus standard therapy over 7 years in patients with systemic lupus erythematosus. J Rheumatol. 2014 Feb;41(2):300-9. doi: 10.3899/jrheum.121368. Epub 2013 Nov 1. PMID 24187095
- [Derived] Struemper H, Chen C, Cai W. Population pharmacokinetics of belimumab following intravenous administration in patients with systemic lupus erythematosus. J Clin Pharmacol. 2013 Jul;53(7):711-20. doi: 10.1002/jcph.104. Epub 2013 May 16. PMID 23681782
- [Derived] Wallace DJ, Navarra S, Petri MA, Gallacher A, Thomas M, Furie R, Levy RA, van Vollenhoven RF, Cooper S, Zhong ZJ, Freimuth W, Cervera R; BLISS-52 and -76, and LBSL02 Study Groups. Safety profile of belimumab: pooled data from placebo-controlled phase 2 and 3 studies in patients with systemic lupus erythematosus. Lupus. 2013 Feb;22(2):144-54. doi: 10.1177/0961203312469259. Epub 2012 Dec 4. PMID 23213069
- [Derived] Merrill JT, Ginzler EM, Wallace DJ, McKay JD, Lisse JR, Aranow C, Wellborne FR, Burnette M, Condemi J, Zhong ZJ, Pineda L, Klein J, Freimuth WW; LBSL02/99 Study Group. Long-term safety profile of belimumab plus standard therapy in patients with systemic lupus erythematosus. Arthritis Rheum. 2012 Oct;64(10):3364-73. doi: 10.1002/art.34564. PMID 22674457
- [Derived] Jacobi AM, Huang W, Wang T, Freimuth W, Sanz I, Furie R, Mackay M, Aranow C, Diamond B, Davidson A. Effect of long-term belimumab treatment on B cells in systemic lupus erythematosus: extension of a phase II, double-blind, placebo-controlled, dose-ranging study. Arthritis Rheum. 2010 Jan;62(1):201-10. doi: 10.1002/art.27189. PMID 20039404

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Plus SOC: Placebo IV plus standard therapy (SOC) for SLE for 52-week double-blind period of the study.
- Belimumab 1 mg/kg Plus SOC: Belimumab 1 mg/kg IV plus standard therapy (SOC) for SLE for 52-week double-blind period of the study. The 24-week open-label extension period of the study included patients who completed the 52-week double-blind period and opted to continue to receive the same dose in the 24-week open-label extension period of the study.
- Belimumab 4 mg/kg Plus SOC: Belimumab 4 mg/kg IV plus standard therapy (SOC) for SLE for 52-week double-blind period of the study. The 24-week open-label extension period of the study included patients who completed the 52-week double-blind period and opted to continue to receive the same dose in the 24-week open-label extension period of the study.
- Belimumab 10 mg/kg Plus SOC: Belimumab 10 mg/kg IV plus standard therapy (SOC) for SLE for 52-week double-blind period of the study. The 24 week-open label extension period of the study included patients who completed the 52-week double-blind period and opted to continue in the 24-week open-label period of the study and included patients who were originally randomized to the belimumab 10 mg/kg group in the double-blind period, patients who switched to belimumab 10 mg/kg at the investigator's discretion, and former placebo patients.
Period: 52-Week Double-Blind Period
Arm/Group | Placebo Plus SOC | Belimumab 1 mg/kg Plus SOC | Belimumab 4 mg/kg Plus SOC | Belimumab 10 mg/kg Plus SOC
Started | 113 | 114 | 111 | 111
Completed | 93 | 87 | 94 | 90
Not Completed | 20 | 27 | 17 | 21
Not completed — Adverse Event | 5 | 8 | 4 | 8
Not completed — Lack of Efficacy | 1 | 2 | 0 | 1
Not completed — Withdrawal by Subject | 7 | 11 | 7 | 7
Not completed — Physician Decision | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 2 | 2
Not completed — Pregnancy | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 1 | 0
Not completed — Death | 0 | 1 | 0 | 0
Not completed — Lack of Compliance | 6 | 3 | 3 | 3
Period: 24-Week Open-Label Extension Period
Arm/Group | Placebo Plus SOC | Belimumab 1 mg/kg Plus SOC | Belimumab 4 mg/kg Plus SOC | Belimumab 10 mg/kg Plus SOC
Started | 0 (Of 93: 88 switched to 10 mg/kg; 5 elected not to continue in the open-label extension period.) | 19 (Of 87: 65 switched to 10 mg/kg; 3 elected not to continue in the open-label extension period.) | 24 (Of 94: 64 switched to 10 mg/kg; 6 elected not to continue in the open-label extension period.) | 302 (Of 90: 85 continued with 10 mg/kg; 5 elected not to continue in the open-label extension period.)
Completed | 0 | 19 | 23 | 279
Not Completed | 0 | 0 | 1 | 23
Not completed — Adverse Event | 0 | 0 | 1 | 6
Not completed — Lack of Efficacy | 0 | 0 | 0 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 9
Not completed — Pregnancy | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 2
Not completed — Lack of Compliance | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Belimumab 1 mg/kg Plus SOC: Belimumab 1 mg/kg IV plus standard therapy (SOC) for SLE for 52-week double-blind period of the study.
- Belimumab 4 mg/kg Plus SOC: Belimumab 4 mg/kg IV plus standard therapy (SOC) for SLE for 52-week double-blind period of the study.
- Belimumab 10 mg/kg Plus SOC: Belimumab 10 mg/kg IV plus standard therapy (SOC) for SLE for 52-week double-blind period of the study.
- Total: Total of all reporting groups
Arm/Group | Placebo Plus SOC | Belimumab 1 mg/kg Plus SOC | Belimumab 4 mg/kg Plus SOC | Belimumab 10 mg/kg Plus SOC | Total
Number analyzed (Participants) | 113 | 114 | 111 | 111 | 449
Age Continuous [Mean (Standard Deviation); unit: years] | 42.2 (10.9) | 42.0 (11.7) | 42.6 (10.7) | 41.8 (11.7) | 42.2 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102 | 107 | 105 | 105 | 419
  Male | 11 | 7 | 6 | 6 | 30
Region of Enrollment [Number; unit: participants]
  United States | 113 | 113 | 111 | 109 | 446
  Canada | 0 | 1 | 0 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Baseline in Safety of Estrogens in Lupus Erythematosus National Assessment SLE Disease Activity Index (SELENA SLEDAI) Score at Week 24.
Description: SELENA SLEDAI is calculated from 24 individual descriptors; 0 indicates inactive disease and the maximum theoretical score is 105; scores > 20 are rare.
Time Frame: Baseline, 24 weeks
Population: Analysis was performed on a modified intention-to-treat (MITT) population, defined as all patients who were randomized and received at least 1 dose of study agent.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo Plus SOC | Belimumab 1 mg/kg Plus SOC | Belimumab 4 mg/kg Plus SOC | Belimumab 10 mg/kg Plus SOC
Number analyzed (Participants) | 113 | 114 | 111 | 111
percent change | -17.2 (5.1) | -23.3 (4.4) | -11.3 (5.4) | -23.7 (4.2)
Statistical Analysis 1: Comparison: Placebo Plus SOC vs Belimumab 1 mg/kg Plus SOC; Missing data was handled by using a last observation carried forward (LOCF) imputation. If patient required a protocol-prohibited medication, the SELENA SLEDAI score of the last visit prior to the use of the prohibited medication was used; Test type: Superiority or Other; p = 0.3677, t-test, 2 sided — P-value was not adjusted for multiple testing; Mean Difference (Final Values) = -6.1, 95% CI 2-sided [-19.4 to 7.2]
Statistical Analysis 2: Comparison: Placebo Plus SOC vs Belimumab 4 mg/kg Plus SOC; Missing data was handled by using LOCF imputation. If patient required a protocol-prohibited medication, the SELENA SLEDAI score of the last visit prior to the use of the prohibited medication was used; Test type: Superiority or Other; p = 0.4244, t-test, 2 sided — P-value was not adjusted for multiple testing; Mean Difference (Final Values) = 5.9, 95% CI 2-sided [-8.7 to 20.6]
Statistical Analysis 3: Comparison: Placebo Plus SOC vs Belimumab 10 mg/kg Plus SOC; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.3296, t-test, 2 sided — P-value was not adjusted for multiple testing; Mean Difference (Final Values) = -6.5, 95% CI 2-sided [-19.6 to 6.6]

2. Primary Outcome: Time to First Mild/Moderate or Severe SLE Flare (SLE Flare Index)
Description: The SLE Flare Index categorized SLE flare as "mild or moderate" or "severe" based on 5 variables: 1) change in SELENA SLEDAI score from the most recent assessment to current, 2) change in signs or symptoms of disease activity, 3) change in prednisone dosage, 4) use of new medications for disease activity or hospitalization, and 5) change in Physician's Global Assessment score, a visual analog scale scored from 0 to 3 (1=mild, 2=moderate, 3=severe).
Time Frame: 0 to 52 weeks
Population: Analysis was performed on a MITT population, defined as all patients who were randomized and received at least 1 dose of study agent.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Placebo Plus SOC | Belimumab 1 mg/kg Plus SOC | Belimumab 4 mg/kg Plus SOC | Belimumab 10 mg/kg Plus SOC
Number analyzed (Participants) | 113 | 114 | 111 | 111
days | 83 [42 to 140] | 68 [39 to 146] | 61 [29 to 147] | 70 [29 to 154]
Statistical Analysis 1: Comparison: Placebo Plus SOC vs Belimumab 1 mg/kg Plus SOC; Patients who required protocol-prohibited medications were considered to have a flare on the date the prohibited medication was started or date of the first flare, whichever came first. Patients who withdrew from the study for reasons other than SLE disease manifestations or hospitalization related to SLE or who missed 2 or more consecutive visits were censored at the time of the last assessment; Test type: Superiority or Other; p = 0.6423, Log Rank — P-value was not adjusted for multiple testing
Statistical Analysis 2: Comparison: Placebo Plus SOC vs Belimumab 4 mg/kg Plus SOC; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.8536, Log Rank — P-value was not adjusted for multiple testing
Statistical Analysis 3: Comparison: Placebo Plus SOC vs Belimumab 10 mg/kg Plus SOC; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.9705, Log Rank — P-value was not adjusted for multiple testing

3. Secondary Outcome: Percentage Change From Baseline in SELENA SLEDAI Score at Week 52
Description: as for outcome 1
Time Frame: Baseline, 52 weeks
Population: as for outcome 2
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo Plus SOC | Belimumab 1 mg/kg Plus SOC | Belimumab 4 mg/kg Plus SOC | Belimumab 10 mg/kg Plus SOC
Number analyzed (Participants) | 113 | 114 | 111 | 111
percent change | -20.6 (5.2) | -29.7 (4.3) | -23.9 (7.3) | -27.9 (5.5)
Statistical Analysis 1: Comparison: Placebo Plus SOC vs Belimumab 1 mg/kg Plus SOC; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.1763, t-test, 2 sided — P-value was not adjusted for multiple testing; Mean Difference (Final Values) = -9.1, 95% CI 2-sided [-22.4 to 4.1]
Statistical Analysis 2: Comparison: Placebo Plus SOC vs Belimumab 4 mg/kg Plus SOC; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.7112, t-test, 2 sided — P-value was not adjusted for multiple testing; Mean Difference (Final Values) = -3.3, 95% CI 2-sided [-20.9 to 14.3]
Statistical Analysis 3: Comparison: Placebo Plus SOC vs Belimumab 10 mg/kg Plus SOC; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.3320, t-test, 2 sided — P-value was not adjusted for multiple testing; Mean Difference (Final Values) = -7.4, 95% CI 2-sided [-22.2 to 7.5]

4. Secondary Outcome: Area Under the Curve (AUC) of SELENA SLEDAI Score at Week 52
Description: SELENA SLEDAI is calculated from 24 individual descriptors; 0 indicates inactive disease and the maximum theoretical score is 105; scores > 20 are rare. The normalized AUC was created as the ratio of the area under the SELENA SLEDAI score curve divided by baseline score.
Time Frame: Baseline and every 4 to 8 weeks through Week 52
Population: as for outcome 2
Measure: Mean (Standard Error); unit: ratio score*days
Arm/Group | Placebo Plus SOC | Belimumab 1 mg/kg Plus SOC | Belimumab 4 mg/kg Plus SOC | Belimumab 10 mg/kg Plus SOC
Number analyzed (Participants) | 113 | 114 | 111 | 111
ratio score*days | 317.3 (14.0) | 288.7 (12.5) | 320.3 (14.0) | 286.9 (13.0)
Statistical Analysis 1: Comparison: Placebo Plus SOC vs Belimumab 1 mg/kg Plus SOC; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.1287, t-test, 2 sided — P-value was not adjusted for multiple testing; Mean Difference (Final Values) = -28.6, 95% CI 2-sided [-65.6 to 8.4]
Statistical Analysis 2: Comparison: Placebo Plus SOC vs Belimumab 4 mg/kg Plus SOC; Missing data was handled by using LOCF imputation; Test type: Superiority or Other; p = 0.8807, t-test, 2 sided — P-value was not adjusted for multiple testing; Mean Difference (Final Values) = 2.98, 95% CI 2-sided [-36.2 to 42.1]
Statistical Analysis 3: Comparison: Placebo Plus SOC vs Belimumab 10 mg/kg Plus SOC; Missing data was handled by using LOCF imputation; Test type: Superiority or Other; p = 0.1131, t-test, 2 sided — P-value was not adjusted for multiple testing; Mean Difference (Final Values) = -30.41, 95% CI 2-sided [-68.1 to 7.3]

5. Secondary Outcome: Percentage Change From Baseline in British Isles Lupus Activity Group (BILAG) Score at Week 52
Description: The BILAG index is a clinical measure of lupus disease activity. BILAG uses a single score for each of the 8 organ domains; range is from severe to no disease (A to E). The global BILAG score is the sum of the numerical scores in the 8 domains assigning A=9, B=3, C=1, D=0, E=0.
Time Frame: Baseline, 52 weeks
Population: as for outcome 2
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo Plus SOC | Belimumab 1 mg/kg Plus SOC | Belimumab 4 mg/kg Plus SOC | Belimumab 10 mg/kg Plus SOC
Number analyzed (Participants) | 113 | 114 | 111 | 111
percent change | -19.1 (4.3) | -20.8 (4.3) | -26.5 (3.4) | -22.0 (4.3)
Statistical Analysis 1: Comparison: Placebo Plus SOC vs Belimumab 1 mg/kg Plus SOC; Missing data for BILAG were handled as described previously for SELENA SLEDAI; Test type: Superiority or Other; p = 0.7823, t-test, 2 sided — P-value was not adjusted for multiple testing; Mean Difference (Final Values) = -1.7, 95% CI 2-sided [-13.8 to 10.4]
Statistical Analysis 2: Comparison: Placebo Plus SOC vs Belimumab 4 mg/kg Plus SOC; Missing data for BILAG were handled as described previously for SELENA SLEDAI; Test type: Superiority or Other; p = 0.1774, t-test, 2 sided — P-value was not adjusted for multiple testing; Mean Difference (Final Values) = -7.4, 95% CI 2-sided [-18.2 to 3.4]
Statistical Analysis 3: Comparison: Placebo Plus SOC vs Belimumab 10 mg/kg Plus SOC; Missing data for BILAG were handled as described previously for SELENA SLEDAI; Test type: Superiority or Other; p = 0.6406, t-test, 2 sided; P-value was not adjusted for multiple testing; Mean Difference (Final Values) = -2.8, 95% CI 2-sided [-14.8 to 9.1]

6. Secondary Outcome: Area Under the Curve (AUC) of BILAG Score at Week 52
Description: The BILAG index is a clinical measure of lupus disease activity. BILAG uses a single score for each of the 8 organ domains; range is from severe to no disease (A to E). The global BILAG score is the sum of the numerical scores in the 8 domains assigning A=9, B=3, C=1, D=0, E=0.The normalized AUC was created as the ratio of the area under the global BILAG score curve divided by baseline score.
Time Frame: Baseline and every 4 to 8 weeks through Week 52
Population: as for outcome 2
Measure: Mean (Standard Error); unit: ratio score*days
Arm/Group | Placebo Plus SOC | Belimumab 1 mg/kg Plus SOC | Belimumab 4 mg/kg Plus SOC | Belimumab 10 mg/kg Plus SOC
Number analyzed (Participants) | 113 | 114 | 111 | 111
ratio score*days | 315.4 (12.3) | 310.6 (12.0) | 300.4 (9.3) | 302.7 (12.3)
Statistical Analysis 1: Comparison: Placebo Plus SOC vs Belimumab 1 mg/kg Plus SOC; Missing data for BILAG were handled as described previously for SELENA SLEDAI; Test type: Superiority or Other; p = 0.7822, t-test, 2 sided — P-value was not adjusted for multiple testing; Mean Difference (Final Values) = -4.8, 95% CI 2-sided [-38.6 to 29.1]
Statistical Analysis 2: Comparison: Placebo Plus SOC vs Belimumab 4 mg/kg Plus SOC; Missing data for BILAG were handled as described previously for SELENA SLEDAI; Test type: Superiority or Other; p = 0.3332, t-test, 2 sided — P-value was not adjusted for multiple testing; Mean Difference (Final Values) = -14.9, 95% CI 2-sided [-45.3 to 15.4]
Statistical Analysis 3: Comparison: Placebo Plus SOC vs Belimumab 10 mg/kg Plus SOC; Missing data for BILAG were handled as described previously for SELENA SLEDAI; Test type: Superiority or Other; p = 0.4660, t-test, 2 sided — P-value was not adjusted for multiple testing; Mean Difference (Final Values) = -12.7, 95% CI 2-sided [-46.9 to 21.5]

7. Secondary Outcome: Time to First Type A/B SLE Flare (as Defined Using BILAG) Over 52 Weeks
Description: SLE flare indicates an increase in SLE disease activity. An SLE flare was a type A or B SLE flare (as defined using BILAG) compared with the previous visit.
Time Frame: 0 to 52 weeks
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Placebo Plus SOC | Belimumab 1 mg/kg Plus SOC | Belimumab 4 mg/kg Plus SOC | Belimumab 10 mg/kg Plus SOC
Number analyzed (Participants) | 113 | 114 | 111 | 111
days | 78 [34 to 138] | 63 [54 to 110] | 84 [51 to 139] | 62 [33 to 108]
Statistical Analysis 1: Comparison: Placebo Plus SOC vs Belimumab 1 mg/kg Plus SOC; Missing data for BILAG were handled as described previously for SELENA SLEDAI (SLE Flare Index); Test type: Superiority or Other; p = 0.5615, Log Rank — P-value was not adjusted for multiple comparisons
Statistical Analysis 2: Comparison: Placebo Plus SOC vs Belimumab 4 mg/kg Plus SOC; Missing data for BILAG were handled as described previously for SELENA SLEDAI (SLE Flare Index); Test type: Superiority or Other; p = 0.7593, Log Rank — P-value was not adjusted for multiple testing
Statistical Analysis 3: Comparison: Placebo Plus SOC vs Belimumab 10 mg/kg Plus SOC; Missing data for BILAG were handled as described previously for SELENA SLEDAI (SLE Flare Index); Test type: Superiority or Other; p = 0.2273, Log Rank — P-value was not adjusted for multiple testing

8. Secondary Outcome: Percentage of Patients With a Reduction in Prednisone Dose
Description: Percentage of patients whose average prednisone dose has been reduced by ≥ 50% and/or has been reduced to ≤ 7.5 mg/day during Weeks 40 through 52 in patients receiving greater than 7.5 mg/day at baseline.
Time Frame: Baseline, weeks 40 to 52
Population: Analysis was performed on a subgroup of the MITT population, which included only patients with baseline prednisone dose > 7.5 mg/day.
Measure: Number; unit: percentatge of particpants
Arm/Group | Placebo Plus SOC | Belimumab 1 mg/kg Plus SOC | Belimumab 4 mg/kg Plus SOC | Belimumab 10 mg/kg Plus SOC
Number analyzed (Participants) | 48 | 40 | 35 | 38
percentatge of particpants | 27.1 | 20.0 | 31.4 | 44.7
Statistical Analysis 1: Comparison: Placebo Plus SOC vs Belimumab 1 mg/kg Plus SOC; Patients who dropped out or had missing data were considered failures; Test type: Superiority or Other; p = 0.4355, Likelihood ratio chi-squared — P-value was not adjusted for multiple testing; percent difference from placebo = -7.1, 95% CI 2-sided [-24.7 to 10.6]
Statistical Analysis 2: Comparison: Placebo Plus SOC vs Belimumab 4 mg/kg Plus SOC; Patients who dropped out or had missing data were considered failures; Test type: Superiority or Other; p = 0.6669, Likelihood ratio chi-squared — P-value was not adjusted for multiple testing; percent difference from placebo = 4.4, 95% CI 2-sided [-15.5 to 24.2]
Statistical Analysis 3: Comparison: Placebo Plus SOC vs Belimumab 10 mg/kg Plus SOC; Patients who dropped out or had missing data were considered failures; Test type: Superiority or Other; p = 0.0882, Likelihood ratio chi-squared — P-value was not adjusted for multiple testing; percent difference from placebo = 17.7, 95% CI 2-sided [-2.5 to 37.9]

9. Other Pre Specified Outcome: Adverse Events (AE) Overview
Description: Includes AEs reported in patients from the first dose of study agent throughout the study up to the Week 76/exit visit or 8 weeks following the last dose of study agent for patients who withdrew from this study or decided not to participate in the optional continuation protocol (LBSL99/NCT00583362).
Time Frame: Up to 84 weeks
Measure: Number; unit: percentage of participants
Groups:
- Open-Label Extension Period: All Active: Includes all patients who completed the 52-week double-blind period and opted to continue in a 24-week open-label extension period. Belimumab patients received the same dose or were switched to belimumab 10 mg/kg at the investigator's discretion and former placebo patients received belimumab 10 mg/kg. AE onset may be during the extension phase or continuing from the double-blind period.
Arm/Group | Placebo Plus SOC | Belimumab 1 mg/kg Plus SOC | Belimumab 4 mg/kg Plus SOC | Belimumab 10 mg/kg Plus SOC | Open-Label Extension Period: All Active
Number analyzed (Participants) | 113 | 114 | 111 | 111 | 345
percentage of participants
  Percent of patients with at least 1 AE | 97.3 | 97.4 | 96.4 | 97.3 | 96.2
  Percent of patients with at least 1 SAE | 19.5 | 18.4 | 13.5 | 16.2 | 9.6
  Percent of patients with an AE resulting in death | 0 | 0.9 | 0 | 0.9 | 0

ADVERSE EVENTS:
Time Frame: Up to 84 weeks
Description: Includes AEs reported in patients from the first dose of study agent throughout the study up to the Week 76/exit visit or 8 weeks following the last dose of study agent for patients who withdrew from this study or decided not to participate in the optional continuation protocol (LBSL99/NCT00583362).
Groups:
- Open-label Extension Period: All Active: Includes all patients who completed the 52-week double-blind period and opted to continue in a 24-week open-label extension period. Belimumab patients received the same dose or were switched to 10 mg/kg at investigator discretion and former placebo patients received belimumab 10 mg/kg. AE onset may be during the extension phase or continuing from the double-blind period.
Arm/Group | Placebo Plus SOC | Belimumab 1 mg/kg Plus SOC | Belimumab 4 mg/kg Plus SOC | Belimumab 10 mg/kg Plus SOC | Open-label Extension Period: All Active
Serious Adverse Events (participants affected / at risk) | 22/113 | 21/114 | 15/111 | 18/111 | 33/345
Other Adverse Events (participants affected / at risk) | 103/113 | 107/114 | 100/111 | 105/111 | 312/345
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Plus SOC (N=113) | Belimumab 1 mg/kg Plus SOC (N=114) | Belimumab 4 mg/kg Plus SOC (N=111) | Belimumab 10 mg/kg Plus SOC (N=111) | Open-label Extension Period: All Active (N=345)
Aplastic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Haemolysis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 1 | 0 | 0 | 0
Pericarditis lupus (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Pleuropericarditis (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Appendicitis noninfective (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gastroduodenitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gastroenteritis noninfectious (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Rectocele (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Adhesion (General disorders) | 1 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 2 | 1 | 0 | 1 | 3
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 2 | 0 | 0
Hepatotoxicity (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Anal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Bronchitis acute (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 2 | 1 | 0 | 1
Clostridium colitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Furuncle (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Lobar pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 2 | 1 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Septic arthritis streptobacillus (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Streptococcal bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Viral infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0
West Nile viral infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Wound infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Seroma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Haematocrit decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Pulmonary function test decreased (Investigations) | 1 | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Spondylosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Metastases to bone marrow (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Cauda equina syndrome (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Grand mal convulsion (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Simple partial seizures (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 2 | 1 | 1 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1 | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0
Completed suicide (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Cystocele (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Glomerulonephritis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Lupus nephritis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0 | 2 | 3
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 1
Menometrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 1
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Vulvar dysplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Chronic obstructive airways disease exacerbated (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 2
Dyspnoea exacerbated (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Angioneurotic oedema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Systemic lupus erythematosus rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Post procedural drainage (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
Arteriosclerosis (Vascular disorders) | 0 | 1 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 1
Hypertensive crisis (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Vasculitis (Vascular disorders) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Plus SOC (N=113) | Belimumab 1 mg/kg Plus SOC (N=114) | Belimumab 4 mg/kg Plus SOC (N=111) | Belimumab 10 mg/kg Plus SOC (N=111) | Open-label Extension Period: All Active (N=345)
Anaemia (Blood and lymphatic system disorders) | 3 | 5 | 7 | 2 | 19
Leukopenia (Blood and lymphatic system disorders) | 5 | 4 | 6 | 9 | 12
Lymphadenopathy (Blood and lymphatic system disorders) | 5 | 2 | 5 | 6 | 5
Abdominal pain (Gastrointestinal disorders) | 9 | 6 | 4 | 4 | 8
Constipation (Gastrointestinal disorders) | 6 | 3 | 4 | 4 | 9
Diarrhoea (Gastrointestinal disorders) | 19 | 19 | 23 | 17 | 34
Dyspepsia (Gastrointestinal disorders) | 8 | 3 | 5 | 7 | 7
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 | 11 | 5 | 7 | 26
Mouth ulceration (Gastrointestinal disorders) | 11 | 9 | 12 | 17 | 18
Nausea (Gastrointestinal disorders) | 27 | 31 | 22 | 33 | 39
Vomiting (Gastrointestinal disorders) | 13 | 14 | 15 | 9 | 15
Fatigue (General disorders) | 34 | 27 | 33 | 27 | 72
Infusion site reaction (General disorders) | 6 | 3 | 12 | 2 | 2
Non-cardiac chest pain (General disorders) | 9 | 6 | 6 | 6 | 9
Oedema peripheral (General disorders) | 13 | 15 | 18 | 15 | 41
Pain (General disorders) | 3 | 1 | 6 | 5 | 12
Pyrexia (General disorders) | 14 | 13 | 17 | 15 | 18
Bronchitis (Infections and infestations) | 7 | 5 | 11 | 14 | 23
Gastroenteritis viral (Infections and infestations) | 4 | 6 | 5 | 4 | 6
Influenza (Infections and infestations) | 8 | 6 | 11 | 7 | 7
Sinusitis (Infections and infestations) | 21 | 11 | 15 | 17 | 34
Upper respiratory tract infection (Infections and infestations) | 33 | 36 | 36 | 29 | 58
Urinary tract infection (Infections and infestations) | 18 | 16 | 18 | 20 | 33
Vaginal mycosis (Infections and infestations) | 8 | 3 | 8 | 4 | 10
Viral infection (Infections and infestations) | 5 | 3 | 8 | 0 | 2
Viral upper respiratory tract infection (Infections and infestations) | 5 | 5 | 6 | 5 | 10
Contusion (Injury, poisoning and procedural complications) | 7 | 10 | 7 | 6 | 12
Creatinine renal clearance decreased (Investigations) | 4 | 5 | 8 | 5 | 8
Weight decreased (Investigations) | 6 | 6 | 5 | 5 | 17
Weight increased (Investigations) | 8 | 6 | 8 | 7 | 28
Decreased appetite (Metabolism and nutrition disorders) | 2 | 6 | 0 | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 42 | 41 | 37 | 41 | 102
Arthritis (Musculoskeletal and connective tissue disorders) | 18 | 16 | 21 | 18 | 47
Back pain (Musculoskeletal and connective tissue disorders) | 16 | 15 | 15 | 16 | 42
Bursitis (Musculoskeletal and connective tissue disorders) | 2 | 6 | 6 | 4 | 7
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 4 | 2 | 5 | 6 | 12
Joint swelling (Musculoskeletal and connective tissue disorders) | 10 | 9 | 11 | 7 | 14
Myalgia (Musculoskeletal and connective tissue disorders) | 14 | 15 | 10 | 15 | 28
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 | 14 | 13 | 10 | 34
SLE arthritis (Musculoskeletal and connective tissue disorders) | 6 | 5 | 2 | 9 | 4
Synovitis (Musculoskeletal and connective tissue disorders) | 4 | 4 | 6 | 6 | 8
Tendonitis (Musculoskeletal and connective tissue disorders) | 3 | 2 | 4 | 8 | 8
Dizziness (Nervous system disorders) | 8 | 8 | 12 | 6 | 10
Headache (Nervous system disorders) | 27 | 29 | 31 | 35 | 50
Hypoaesthesia (Nervous system disorders) | 3 | 4 | 5 | 6 | 13
Migraine (Nervous system disorders) | 11 | 11 | 6 | 15 | 19
Paraesthesia (Nervous system disorders) | 1 | 7 | 3 | 1 | 4
Sinus headache (Nervous system disorders) | 6 | 1 | 0 | 2 | 3
Anxiety (Psychiatric disorders) | 6 | 6 | 8 | 3 | 19
Depression (Psychiatric disorders) | 9 | 16 | 12 | 10 | 31
Insomnia (Psychiatric disorders) | 10 | 5 | 5 | 9 | 35
Haematuria (Renal and urinary disorders) | 3 | 3 | 4 | 7 | 5
Proteinuria (Renal and urinary disorders) | 6 | 6 | 7 | 4 | 17
Pyuria (Renal and urinary disorders) | 1 | 6 | 4 | 3 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 13 | 8 | 13 | 25
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 3 | 8 | 9 | 17
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 0 | 7 | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 9 | 6 | 3 | 2 | 7
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 2 | 6 | 2 | 6 | 5
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 7 | 5 | 2 | 5
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 9 | 5 | 4 | 2 | 7
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 7 | 6 | 6 | 5 | 7
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 8 | 4 | 1 | 3 | 6
Alopecia (Skin and subcutaneous tissue disorders) | 13 | 10 | 9 | 11 | 24
Erythema (Skin and subcutaneous tissue disorders) | 4 | 6 | 10 | 3 | 12
Pruritus (Skin and subcutaneous tissue disorders) | 8 | 5 | 5 | 8 | 13
Rash (Skin and subcutaneous tissue disorders) | 12 | 16 | 17 | 8 | 25
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 9 | 3 | 7 | 6 | 13
Systemic lupus erythematosus rash (Skin and subcutaneous tissue disorders) | 5 | 2 | 4 | 6 | 12
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 5 | 6 | 3 | 6
Hypertension (Vascular disorders) | 5 | 6 | 5 | 13 | 25
Raynaud's phenomenon (Vascular disorders) | 4 | 6 | 4 | 4 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.